CLINICAL TRIAL: NCT00296764
Title: Angelman Syndrome Natural History Study
Brief Title: Characterization of Angelman Syndrome
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Rady Children's Hospital, San Diego (Other); Baylor College of Medicine (Other); Greenwood Genetic Center (Other); Children's Hospital Medical Center, Cincinnati (Other); Vanderbilt University Medical Center (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Wen-Hann Tan, Site PI (Lead PI: Lynne M. Bird, MD - Univ. of California, San Diego), Boston Children's Hospital
Other Study IDs: RDCRN 5203; U54RR019478 (NIH)
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Angelman Syndrome
Keywords: Developmental Disorders
MeSH Terms: conditions — Angelman Syndrome; Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and cheek swab samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Angelman Syndrome (AS) is a developmental disorder that is caused by a deficiency of a maternally transmitted gene. It is inherited at birth, and affects movement, speech, and social demeanor. This study will gain a better understanding of the disease progression and clinical features of AS by observing children with AS over an extended period of time.

DETAILED DESCRIPTION:
AS is a developmental disorder that affects movement, speech, and social demeanor. The disorder is caused by a deficiency of a maternally transmitted gene and is inherited at birth. Children with AS, however, are often not diagnosed until they are between 3 and 7 years old. Symptoms of AS may include, but are not limited to, functionally severe developmental delay; speech impairments; movement or balance problems; and behavioral uniqueness, including any combination of frequent laughter or smiling, apparent happy demeanor, easily excitable personality, hand flapping movements, and short attention span. There are four molecular variations of AS, but past clinical studies have been inconsistent in highlighting the phenotypic differences between them. This study will gain a better understanding of the disease progression and clinical features of AS by observing children with AS over a period of 5 to 10 years. The study will also attempt to establish genotype-phenotype correlations, which might aid in future clinical care of AS patients.

Participation in this observational study will be limited to current or future patients at one of the five study sites. A clinical evaluation will be performed at baseline, including a general patient history, physical and neurological examinations, a nutritional assessment, neuro-imaging, electroencephalography, laboratory testing, and neurodevelopmental testing. A blood sample or mucosal sample will also be taken at baseline to acquire DNA for potential genetic testing. All assessments except the neuro-imaging, electroencephalography, and blood sampling will be repeated at yearly study visits for as long as funding can be secured. In addition, participants will be photographed and perhaps videotaped on a yearly basis in order to document clinical phenotypes and any neurologic abnormalities. Participants may be followed-up for a total of 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Molecular diagnosis of Angelman syndrome OR
2. Meets all major diagnostic criteria for Angelman Syndrome and 3 of the 6 minor criteria:

Major Criteria:

* Functionally severe developmental delay
* Speech impairment; none or minimal words used
* Movement or balance disorder
* Behavioral uniqueness, frequent laughs/smiling, excitable personality, hand flapping, short attention span

Minor Criteria:

* Deceleration in head circumference growth (post-natal)
* Seizures (myoclonic, absence, drop, tonic-clonic)
* Abnormal EEG (with patterns suggestive of AS, or hypsarrhythmia)
* Sleep disturbance
* Attraction to or fascination with water
* Drooling

Exclusion Criteria:

* Does not meet diagnostic criteria for Angelman Syndrome
* Other medical or genetic disorders (except autism)
* Born extremely premature

Ages: 1 Day to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Angelman syndrome (molecular or clinical diagnosis) between the ages of 1 day and 60 years.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
medical morbidity | annually
  to characterize the medical problems associated with Angelman syndrome, and to determine the relative prevalence of those problems in the different molecular subclasses of Angelman syndrome
developmental progress | annually
  Assess with a variety of neuropsychological instruments, including Bayley Scales of Infant Development, Vineland Adaptive Behavior Scales, Preschool Language Scale

SECONDARY OUTCOMES:
autism | annually
  Evaluate for autism spectrum disorder using Autism Diagnostic Observation Schedule and Autism Diagnostic Interview-Revised

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A. Bacino, MD, Principal Investigator — Baylor College of Medicine, Department of Molecular and Human Genetics; Lynne Bird, MD, Study Chair — Rady Childrens Hospital San Diego, UCSD Dept of Pediatrics; Steven A. Skinner, MD, Principal Investigator — Greenwood Genetic Center; Wen-Hann Tan, BMBS, Principal Investigator — Boston Children's Hospital; Logan K Wink, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Sarika Peters, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (6):
- United States (6):
  - Rady Children's Hospital San Diego, San Diego, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varela MC, Kok F, Otto PA, Koiffmann CP. Phenotypic variability in Angelman syndrome: comparison among different deletion classes and between deletion and UPD subjects. Eur J Hum Genet. 2004 Dec;12(12):987-92. doi: 10.1038/sj.ejhg.5201264. PMID 15470370
- [Background] Peters SU, Beaudet AL, Madduri N, Bacino CA. Autism in Angelman syndrome: implications for autism research. Clin Genet. 2004 Dec;66(6):530-6. doi: 10.1111/j.1399-0004.2004.00362.x. PMID 15521981
- [Background] Locke DP, Segraves R, Nicholls RD, Schwartz S, Pinkel D, Albertson DG, Eichler EE. BAC microarray analysis of 15q11-q13 rearrangements and the impact of segmental duplications. J Med Genet. 2004 Mar;41(3):175-82. doi: 10.1136/jmg.2003.013813. PMID 14985376
- [Background] Smith JC. Angelman syndrome: evolution of the phenotype in adolescents and adults. Dev Med Child Neurol. 2001 Jul;43(7):476-80. doi: 10.1017/s0012162201000871. PMID 11463179
- [Background] Williams CA, Lossie A, Driscoll D; R.C. Phillips Unit. Angelman syndrome: mimicking conditions and phenotypes. Am J Med Genet. 2001 Jun 1;101(1):59-64. doi: 10.1002/ajmg.1316. PMID 11343340
- [Derived] Frohlich J, Chiang JN, Mediano PAM, Nespeca M, Saravanapandian V, Toker D, Dell'Italia J, Hipp JF, Jeste SS, Chu CJ, Bird LM, Monti MM. Neural complexity is a common denominator of human consciousness across diverse regimes of cortical dynamics. Commun Biol. 2022 Dec 15;5(1):1374. doi: 10.1038/s42003-022-04331-7. PMID 36522453
- [Derived] Keute M, Miller MT, Krishnan ML, Sadhwani A, Chamberlain S, Thibert RL, Tan WH, Bird LM, Hipp JF. Angelman syndrome genotypes manifest varying degrees of clinical severity and developmental impairment. Mol Psychiatry. 2021 Jul;26(7):3625-3633. doi: 10.1038/s41380-020-0858-6. Epub 2020 Aug 13. PMID 32792659
- [Derived] Frohlich J, Miller MT, Bird LM, Garces P, Purtell H, Hoener MC, Philpot BD, Sidorov MS, Tan WH, Hernandez MC, Rotenberg A, Jeste SS, Krishnan M, Khwaja O, Hipp JF. Electrophysiological Phenotype in Angelman Syndrome Differs Between Genotypes. Biol Psychiatry. 2019 May 1;85(9):752-759. doi: 10.1016/j.biopsych.2019.01.008. Epub 2019 Jan 19. PMID 30826071
- [Derived] Killian JT, Lane JB, Cutter GR, Skinner SA, Kaufmann WE, Tarquinio DC, Glaze DG, Motil KJ, Neul JL, Percy AK. Pubertal development in Rett syndrome deviates from typical females. Pediatr Neurol. 2014 Dec;51(6):769-75. doi: 10.1016/j.pediatrneurol.2014.08.013. Epub 2014 Aug 29. PMID 25283752
- [Derived] Neul JL, Lane JB, Lee HS, Geerts S, Barrish JO, Annese F, Baggett LM, Barnes K, Skinner SA, Motil KJ, Glaze DG, Kaufmann WE, Percy AK. Developmental delay in Rett syndrome: data from the natural history study. J Neurodev Disord. 2014;6(1):20. doi: 10.1186/1866-1955-6-20. Epub 2014 Jul 22. PMID 25071871